CLINICAL TRIAL: NCT05310318
Title: Surgical and Reproductive Results of Fertility-sparing Treatment for Low-grade Endometrial Stromal Sarcoma: A Retrospective Cohort Study
Brief Title: Prognosis of Low-grade Endometrial Stromal Sarcoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: SOUM-2
Record Dates: First submitted 2022-03-26; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Low Grade Endometrial Stromal Sarcoma of Uterus (Diagnosis); Fertility-sparing Surgery; Survival Outcomes; Fertility Outcomes; Recurrence; Hormone Therapy; Adjuvant Therapy
MeSH Terms: conditions — Endometrial Stromal Tumors; Disease; Recurrence | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgical treatment with and without fertility-sparing procedures — Patients accepted surgeries for LGESS and relevant adjuvant therapy if indicated.
  Other Names: Adjuvant therapy after surgery

SUMMARY:
This study is to investigate the survival outcomes and fertility outcomes in patients with uterine low-grade endometrial stromal sarcoma (LGESS) treated in Peking Union Medical College Hospital. All primary and recurrent LGESS patients will be enrolled. The study will collect retrospectively data consisting of epidemiological characteristics, surgical, medical treatment and adjuvant therapy. Details about recurrence, mortality, pregnancy and obstetrical outcomes are also followed as primary endpoints. Fertility-sparing procedures, including uterine-sparing and ovary-sparing surgeries will be recorded specifically.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Confirmed of LGESS
* Acceptance of surgical treatment for LGESS
* With detailed follow-up outcomes

Exclusion Criteria:

- Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients accepted surgical treatment with and without fertility-sparing procedures for uterine low-grade endometrial stromal sarcoma.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-03-26 (Actual); Primary Completion 2024-03-26 (Estimated); Study Completion 2025-03-26 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | One year
  Progression-free survival after surgery
Overall survival | One year
  Overall survival after surgery
Pregnancy rate | One year
  Pregnancy rate after surgery in patients with fertility-sparing patients

SECONDARY OUTCOMES:
Miscarriage rate | One year
  Miscarriage rate after surgery in patients with fertility-sparing patients
Full-term pregnancy rate | One year
  Full-term pregnancy rate after surgery in patients with fertility-sparing patients

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China